CLINICAL TRIAL: NCT04044729
Title: Exploring the Mechanisms Underlying the Analgesic Properties of Cannabidiol Using Magnetic Resonance Spectroscopy
Brief Title: Mechanisms of CBD for Chronic Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Deborah Yurgelun-Todd, Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00124865
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Active Comparator): Drug: Cannabidiol An oral dose of Cannabidiol (CBD) will be given once a day for five day with pain ratings taken before and after each dose every day.
  Other Names:
  CBD
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Drug: Placebos An oral placebo will be given once a day for five day with pain ratings taken before and after each dose every day.
  Other Names:
  placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — 500mg dose, suspended in medical grade olive oil and then mixed into chocolate pudding
  Arms: Cannabidiol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a study designed to examine the neurochemical mechanisms associated with Cannabidiol (CBD) versus placebo for chronic non-cancer pain.

DETAILED DESCRIPTION:
The aim of this trial is to examine the neurochemical mechanisms associated with Cannabidiol (CBD) versus placebo for chronic non-cancer pain. Participants will include individuals with chronic pain, who will be randomized into one of two intervention conditions: low THC/high CBD or placebo. In addition to receiving CBD or placebo, participants also will complete symptom assessments of chronic pain data (intensity, quality, interference/disability) throughout the study. These measures will be gathered prior to and following the fifth doses (dosing will occur once per day for five days) of CBD or placebo. A secondary objective will be to examine the association between clinical and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 yrs.
* Chronic musculoskeletal and joint pain for at least 3 months or longer.
* Participants must live within a 60 mile radius of Salt Lake City, Utah to be eligible.

Exclusion Criteria:

* Current or past neurological illness.
* Substance abuse or dependence within the prior 90 days.
* Contraindication to brain MRI.
* Type I and type II diabetes.
* Unstable medical conditions.
* Consumption of more than 2 drinks of alcohol per night.
* Current pregnancy or planning to become pregnant or breastfeeding.
* History of seizures or head trauma at PI discretion.
* Active or history of major mental illness
* Use of opioid medications in the past 30 days.
* LFT results 3 times greater than the upper limit of normal at the screening.
* Participants may be excluded if the PI feels they do not meet safety criteria.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Neurochemical Brain Changes | 5 Days
  Participants will undergo MRS scanning to assess neurochemical shifts from the baseline visit (day 1) to the visit five (day 5) in order to determine whether CBD, or Placebo will result in changes to neurochemical ratios in select brain regions. Neurotransmitter levels such as BABA and N-Acetylaspartate will be collected and compared pre and post study drug administration.

SECONDARY OUTCOMES:
Pain Improvement | 7 Days
  Using baseline assessment measures gathered at visit 0 (Screening), assessments collected at visits 1-5 and follow-up will be used to determine whether the administration of CBD or placebo will improve pain relief in individuals with chronic pain. We will measure pain intensity with a visual analog scale from (0-10) with 10 being the worst pain imaginable. We will also measure Objective pain thresholds with a pressure algometer. This is a device that applies pressure to the participants finger until they say stop. The pressure range is 0-50 foot pounds of force.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are still deciding on if and what IPD will be shared and the details involved. The investigators will update when a plan is in place.